CLINICAL TRIAL: NCT01384292
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of NKTR-118 in Relieving Opioid-Induced Constipation (OIC) in Patients With Cancer-Related Pain
Brief Title: Assessment of Efficacy and Safety in Relieving Opioid-induced Constipation in Patients With Cancer-related Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped early due to recruitment challenges
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3820C00006; 2011-001985-16
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Opioid-Induced Constipation
Keywords: Cancer-Related Pain; Opioid-Induced Constipation; OIC
MeSH Terms: conditions — Opioid-Induced Constipation; Cancer Pain | interventions — naloxegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (part A and B) (Experimental): Oral treatment
  Interventions: Drug: NKTR-118
- 2 (part A and B) (Experimental): Oral treatment
  Interventions: Drug: NKTR-118
- 3 (part A only) (Placebo Comparator): Oral treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NKTR-118 — 12.5 mg oral tablet once daily
  Arms: 1 (part A and B)
Drug: NKTR-118 — 25 mg oral tablet once daily
  Arms: 2 (part A and B)
Drug: Placebo — Oral treatment
  Arms: 3 (part A only)

SUMMARY:
The purpose of this study is to compare the effect of NKTR-118 with placebo in the treatment of opioid-induced constipation (OIC) in patients with cancer-related pain, including those patients that have inadequate response to laxative therapy (LIR).

The study consists of 2 parts; A initial 4-week treatment period (part A) and then a 12 week extension with active treatment (part B).

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any study-specific procedures.
* Men and women aged 18 or older.
* Histologically or cytologically confirmed neoplasm causing pain and requiring management with opioids.
* Self-reported active symptoms of OIC at screening (<3 RFBMs/week and experiencing >1 reported symptom of hard/lumpy stools, straining, or sensation of incomplete evacuation/anorectal obstruction in at least 25% of BMs over the previous 4 weeks); and Documented confirmed OIC (<3 RFBMs/week on average aver the 2-week OIC confirmation period.
* Receiving a stable maintenance opioid regimen consisting of a total daily dose of >30 mg of oral morphine, or equianalgesic amount(s) of 1 or more opioid therapies for a minimum of 4 weeks prior to screening for cancer-related pain with no anticipated change in opioid dose requirement over the proposed study period as a result of disease progression.

Exclusion Criteria:

* Patients receiving Opioid regimen for treatment of pain other than related to cancer.
* Any condition that may have affected the permeability of the blood-brain barrier, eg, known brain metastases, meningeal metastases, brain injury, multiple sclerosis, recent brain injury, uncontrolled epilepsy.
* Patients with cancer-related pain due to ovarian cancer, leukaemia, or lymphoma are excluded. Patients with multiple myeloma will be allowed.
* Patients requiring radiation therapy between the diaphragm and pelvis 4 weeks prior to Visit 1 (screening) and/or during Part A of the study are excluded. Any patients with suspected clinically relevant radiation-induced injury of small or large intestine are excluded.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (140):
- United States (81):
  - Research Site, Huntsville, Alabama
  - Research Site, Casa Grande, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Fort Smith, Arkansas
  - Research Site, Hot Springs, Arkansas
  - Research Site, North Little Rock, Arkansas
  - Research Site, Encino, California
  - Research Site, Fountain Valley, California
  - Research Site, Gilroy, California
  - Research Site, Laguna Hills, California
  - Research Site, Montebello, California
  - Research Site, Orange, California
  - Research Site, Riverside, California
  - Research Site, San Bernardino, California
  - Research Site, Aurora, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Baypines, Florida
  - Research Site, Boynton Beach, Florida
  - Research Site, Celebration, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Naples, Florida
  - Research Site, Plantation, Florida
  - Research Site, Tavares, Florida
  - Research Site, Albany, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Riverdale, Georgia
  - Research Site, Roswell, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Chicago, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Anderson, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Owensboro, Kentucky
  - Research Site, Lafayette, Louisiana
  - Research Site, Elkridge, Maryland
  - Research Site, Hollywood, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Fairhaven, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Southaven, Mississippi
  - Research Site, Jefferson City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Toms River, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Great Neck, New York
  - Research Site, Syracuse, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Flat Rock, North Carolina
  - Research Site, Morrisville, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Bismarck, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Beavercreek, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Middleton, Ohio
  - Research Site, Danville, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Beaumont, Texas
  - Research Site, Bellaire, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Lubbock, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sugarland, Texas
  - Research Site, Fairfax, Virginia
- Australia (5):
  - Research Site, Broadmeadow, New South Wales
  - Research Site, Frankston, Victoria
  - Research Site, Malvern, Victoria
  - Research Site, Parkville, Victoria
  - Research Site, Fremantle, Western Australia
- Belgium (4):
  - Research Site, Edegem, Belgium
  - Research Site, Mons, Belgium
  - Research Site, Brussels
  - Research Site, Wetteren
- Bulgaria (6):
  - Research Site, Haskovo
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Shumen
  - Research Site, Sofia
  - Research Site, Varna
- Research Site, Zagreb, Croatia
- Czechia (3):
  - Research Site, Benešov
  - Research Site, České Budějovice
  - Research Site, Prague
- Germany (4):
  - Research Site, Hamburg, Hamburg
  - Research Site, Wiesbaden, Hesse
  - Research Site, Berlin, State of Berlin
  - Research Site, Offenbach
- Poland (7):
  - Research Site, Brzozów
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Gliwice
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Research Site, Ponce, Puerto Rico
- Romania (8):
  - Research Site, Craiova, Dolj
  - Research Site, Ploieşti, Prahova
  - Research Site, Baia Mare
  - Research Site, Brasov
  - Research Site, Brăila
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Onești
- Slovakia (4):
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Prešov
- South Africa (7):
  - Research Site, Port Elizabeth, Eastern Cape
  - Research Site, Bloemfontein, Free State
  - Research Site, Benoni, Gauteng
  - Research Site, Pretoria, Gauteng
  - Research Site, Vereeniging, Gauteng
  - Research Site, Durban, Kz-natal
  - Research Site, Goodwood, W Cape
- Spain (3):
  - Research Site, Seville, Andalusia
  - Research Site, A Coruña, Galicia
  - Research Site, Valencia, Valencia
- United Kingdom (6):
  - Research Site, Penarth, CRF
  - Research Site, Norwich, Norfolk
  - Research Site, Guildford, Surrey
  - Research Site, Chippenham, Wilts
  - Research Site, Coventry
  - Research Site, London

REFERENCES:
- See also: Clinical_Study_Report_Synopsis_D3820C00006 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1388&filename=Clinical_Study_Report_Synopsis_D3820C00006.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in Poland, the Czech Republic, and the United States between 29 June 2011 and 20 September 2012. Due to recruitment challenges, enrollment to this study was stopped early and no new patients had been screened as of 20 April 2012. Fourteen patients were randomized across the 3 treatment groups.
Pre-assignment Details: Part A was 8 weeks: 14-day screening period, 2-week OIC confirmation period, 4-week treatment period. Part B was 14 weeks: 12-week treatment period, 2-week follow-up period. Part B was optional for eligible patients completing Part A. NKTR-118 patients from Part A remained on the same NKTR-118 dose, while placebo patients received NKTR-118 25 mg.
Groups:
- NKTR-118 12.5 mg: NKTR-118 12.5 mg, oral treatment
- NKTR-118 25 mg: NKTR-118 25 mg, oral treatment
- Placebo: Placebo, oral treatment
Period: Part A
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Started | 5 | 5 | 4
Completed | 5 | 5 | 4
Not Completed | 0 | 0 | 0
Period: Part B
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Started | 3 | 6 | 0
Completed | 2 | 6 | 0
Not Completed | 1 | 0 | 0
Not completed — Severe non-compliance to protocol | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.8 (9.20) | 53.8 (11.69) | 52.5 (4.93) | 54.1 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 10
  Male | 2 | 1 | 1 | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 5 | 3 | 3 | 11
  Black or African American | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Response (Responder/Non-responder) to Study Drug
Description: Response (responder/non-responder) to study drug, where a responder was defined as having at least 3 rescue-free bowel movements (RFBMs) per week during the 4-week Part A treatment period, with at least 1 RFBM per week increase over baseline for at least 3 out of 4 weeks. An RFBM was defined as a bowel movement (BM) without rescue laxatives in the previous 24 hours.
Time Frame: Baseline to Week 4
Population: All randomized patients
Measure: Number; unit: Participants
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 5 | 5 | 4
Participants | 4 | 3 | 2

ADVERSE EVENTS:
Groups:
- NKTR-118 12.5 mg - Part A: Part A NKTR-118 12.5 mg, oral treatment
- NKTR-118 25 mg - Part A: Part A NKTR-118 25 mg, oral treatment
- Placebo - Part A: Part A Placebo, oral treatment
- NKTR-118 12.5 mg - Part B: Part B NKTR-118 12.5 mg, oral treatment
- NKTR-118 25 mg - Part B: Part B NKTR-118 25 mg, oral treatment
Arm/Group | NKTR-118 12.5 mg - Part A | NKTR-118 25 mg - Part A | Placebo - Part A | NKTR-118 12.5 mg - Part B | NKTR-118 25 mg - Part B
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/4 | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 4/5 | 3/5 | 3/4 | 1/3 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKTR-118 12.5 mg - Part A (N=5) | NKTR-118 25 mg - Part A (N=5) | Placebo - Part A (N=4) | NKTR-118 12.5 mg - Part B (N=3) | NKTR-118 25 mg - Part B (N=6)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to recruitment challenges, enrollment was stopped early. 14 patients were randomized (<5% of planned number), thus, there was insufficient data to perform the protocol-specified statistical analyses. Secondary outcome measures are not reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days